CLINICAL TRIAL: NCT03558802
Title: Exploring Pelvic Floor Signs and Symptoms in Community Dwelling Women and Men: a Mixed-method Study
Brief Title: Pelvic Floor Signs and Symptoms in Women and Men
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Grietje E Knol-de Vries, PhD, coordinating investigator Postdoc researcher, University Medical Center Groningen
Other Study IDs: NL67503.042.18; 201800687 (Registry Identifier: Research Register University Medical Center Groningen UMCG)
Record Dates: First submitted 2018-05-15; First posted 2018-06-15 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — questionnaire

SUMMARY:
Rationale: Pelvic floor symptoms (PFS) are prevalent and often impair quality of life. They include micturition problems, defecation problems, pelvic organ prolapse, sexual problems and genito-pelvic pain. The pelvic floor is an anatomical and functional unit, and therefore different PFS may co-occur. However, literature on prevalence of clusters of PFS is scarce. Furthermore, PFS is understudied in the male population and when studies are performed in male subjects, studies do not assess the complete scope of possible PFS.

Objective: To generate a cohort, which provides information on sex- and gender differences in: prevalence and incidence of (clinically relevant clusters of) PFS, risk factors and prognostic factors for PFS, factors that reveal the impact of PFS on daily life, help seeking behavior and use of health care.

Study design: Prospective observational population-based cohort study with follow-up moments after 1 year and 2 years. Data of the questionnaire will be connected to medical record data from the participating general practitioners (GPs). A representative sample of female and male subjects with and without PFS will be invited for a physical examination to assess pelvic floor disorders and muscle function. Furthermore, a subsample of patients will be invited for a qualitative study consisting of semi-structured interviews on healthcare seeking behavior, including barriers and facilitators, preferences and satisfaction.

Study population: female and male subjects, aged ≥16 years of age, from the general population will be included. Exclusion criteria are: terminal disease, or dementia, cognitive impairment or current psychological condition precluding informed consent, not suitable or too ill to participate based on the judgement of the GP.

Main study parameters: To evaluate the sex- and gender difference in prevalence and incidence of (clinically relevant clusters of) PFS, the following primary parameters are assessed: lower urinary tract symptoms, bowel symptoms, urogenital prolapse (females only), sexual functioning, and pain. Secondary study parameters are factors associated with the development of PFS ('risk factors'), factors that predict the course of PFS ('prognostic factors'), factors that reveal the impact of PFS on daily life, help seeking behavior, and health care use (consultations for PFS and consultation frequency, diagnostic tests, diagnoses, treatment, and referrals).

DETAILED DESCRIPTION:
Primary Objective:

To explore sex- and gender differences in:

1. the prevalence of (clinically relevant clusters) of PFS
2. the incidence of (clinically relevant clusters) of PFS

   Secondary Objectives:

   To explore sex- and gender differences in:
3. factors associated with the development of PFS ('risk factors')
4. factors that predict the course of PFS ('prognostic factors')
5. factors that reveal the impact of PFS on daily life
6. help seeking behavior
7. health care use (consultations for PFS and consultation frequency, diagnostic tests, diagnoses, treatment, and referrals) among those who sought care.

Design:

For this study a mixed-methods approach will be used, combining quantitative and qualitative study designs.

The first step is to set-up a prospective population-based cohort study with a 2-year follow-up based on annual self-administered questionnaires. Eligible participants will be invited by general practices in a well-defined region: the municipality of Coevorden.

Electronic medical record data (extracted from the Huisartsen Informatie Systeem, HIS) will be matched with outcomes of the questionnaire, by a trusted third party (TTP).

A sample of female (n=200) and male (n=200) subjects with and without PFS will be invited for physical examination to assess pelvic floor disorders and pelvic floor muscle function (sub study 1).

A sample of patients with PFS will be invited for a qualitative study consisting of a semi-structured interview on help seeking behavior, including barriers and facilitators, preferences and satisfaction (sub study 2).

Procedures:

In the upcoming period before the baseline questionnaire the study will be given attention by flyers/posters in the waiting room of the participating practices and local press.

Eligible persons will receive an information letter, with informed consent form attached, from their GP about the cohort study.

Informed consent:

People can provide informed consent by sending a signed informed consent form to the coordinating investigator using the pre-stamped and self-addressed envelope included.

Subjects will be asked to fill in the informed consent form for

1. participation in the cohort study (i.e. filling in the questionnaire),
2. permission to collect medical GP record data
3. permission to be approached for future sub-studies

   Filling in the questionnaire:

   After providing informed consent, participants will receive an e-mail including the website of the questionnaire and their unique personal code for filling in the questionnaire.

   When subjects have not finished the questionnaire within 2 weeks, they will receive an automatically generated reminder by e-mail. When 1 week after the e-mail reminder, the subject has not finished the questionnaire, a second reminder by SMS will be sent. If a subject will not respond to these reminders, he/she will be considered as nonresponder (baseline) or lost to follow up.

   The questionnaire consists of 11 parts for women and 10 parts for men, with a filling in time of approximately 45-60 minutes. Subjects may interrupt completing the questionnaire and continue it later on. In the online version there will be a button that enables completing the questionnaire in another time (details on the questionnaire can be found in the Methods section of this protocol). The questions in the online questionnaire will have audio support, to stimulate participation and prevent drop-out of participants with low literacy.

   Subjects, who do not have access to the internet can use a laptop of the research team, made available in the local general practice (in a private room). Subjects who indicated that they want to fill in a paper version of the questionnaire will receive a paper version at their home address including a pre-stamped and self-addressed envelope. The paper questionnaires (provided only with the subject identification code) will be entered into the online RoQua system by the coordinating researcher or research assistant.

   In case participants need support with filling in the questionnaires, such support is provided through the research team in the municipality of Coevorden. For this, medical students (males and females) with different native languages will be deployed. Due to the privacy sensitive nature of the study, we actively discourage participants to ask support from their peers or family.

   Invitation and procedure for sub-studies Eligible participants (see information on sub-studies), who provided informed consent for receiving information on sub-studies, will receive a participant information leaflet for the specific sub-study.

   Sub study 1 physical examination When participants (at least 21 years old) want to participate they fill in the reply form and send it to the research team. A member of the research team will schedule an appointment for the physical examination. The participant and a member of the study team will sign informed consent face to face before the start of the physical examination.

   Sub study 2 interview When participants want to participate they fill in the informed consent form and send it to the research team. A member of the research team will schedule an appointment for the interview.

   Follow-up:

   Participants who completed the baseline questionnaire will be invited after 1 year and after 2 years to participate in the follow-up questionnaire rounds.

   Data:

   1. List with potential participants (key file) In order to invite subjects (after informed consent), to send reminders to the subjects, and to eventually connect the questionnaire database with the medical record data, this data file contains information about sex, name, date of birth, address, postal code, place, email-address, and telephone number. Furthermore, preference of way of filling in the questionnaire (online or paper, with or without guidance), and permission to collect medical GP record data, and permission to be approached for future sub-studies will be included in this data file.

   A subject identification code will be made for each subject. This code is not based on patient initials and birth-date. The data file is safeguarded by the coordinating investigator and the research assistant that is part of the research team, and will be stored in a separate place apart from other files, without access from outside. A password will be needed for entering this key file.

   2a. Data file with personal data In order to connect subjects to the questionnaire database, and to send reminders to the subjects, this data file contains information about sex, name, email-address, telephone number and the subject identification number.

   This system with personal data will be filled in by predefined research members (i.e. the coordinating researcher and research assistant of the study) and access to the system is restricted to those predefined research members. Next to a login account, the system is secured by Google Authenticator. The predefined research members have restricted options, such as filling in the personal data and inviting subjects for filling in the questionnaire.

   2b. Questionnaire database RedCap will be used to collect and store data generated from the questionnaires. Data are stored servers under the management of 'het Centrum voor Informatie Technologie (CIT)' of the RuG. The database is not directly accessible for the researcher, but will be made available to the researcher according to the approved Research Data management plan. Data will not be anonymized, but pseudonymized as it is necessary to trace data to an individual subject. This procedure will be performed by a Trusted Third Party (ZorgTTP).

   3. Medical data GPs Medical data will be collected through the electronic medical records (Huisarts Informatie Systeem, HIS) systems used by the different general practices. Data from those HIS systems will be collected via VIPLive and transformed by Calculus/Proigia in order to generate a generic structure of the data. The structured data will then be returned to VIPLive and will be sent to ZorgTTP for pseudomization. The pseudonymized data are sent to the AHON (Academisch Huisarts Ontwikkel Netwerk) database. The time scale for medical record review is 5 years prior to baseline measurement up to the end of follow-up in the cohort.

   4. Research database The different databases (questionnaire database and a subset of the AHON database) can be connected via the unique pseudomization codes provided by ZorgTTP, eventually resulting in a secured research database. This raw data file will be locked for editing after closure of the study. Data cleaning and processing will be executed using syntaxes in program SPSS.

   Monitoring and Quality Assurance:

   As this study is with negligible risks a monitor from the University Medical Center Groningen (UMCG) will monitor the study.

   Statistical analysis:

   Primary study parameter(s):

   To identify distinct classes of patients with clinically relevant clusters of PFS we will perform Latent Class Analyses (LCA). LCA is a type of cluster analysis used to group patients into k number of unique categories, where, within each category patients are most similar to each other regarding PFS, and between the categories patients are most different. The prevalence and incidence of those clinically relevant clusters of PFS will be calculated.

   To explore whether sex- and gender-differences are present, we will perform most of the analyses separately for sex (male and female subjects). The main reason for this is that the questionnaires to measure PFS among women (female subjects) and men (male subjects) are different to each other.

   Secondary study parameter(s):

   Univariate analyses will be performed to assess which parameters will be used in the multivariable regression-analyses. In addition to those univariate parameters, parameters known from literature will be added to the regression models.

   Multivariable regression-analyses will be used to assess which factors are associated with cluster membership. We aim to distinguish factors associated with the development of PFS ('risk factors'), factors that predict the course of PFS ('prognostic factors'), factors that reveal the impact of PFS on daily life, and explore sex and gender differences.

   To determine which factors are potential risk factors, a subsample consisting of participants without PFS at baseline will be selected.

   Multivariable regression-analyses will be used to identify baseline factors that are associated with the development of PFS at follow-up measurements. To determine which factors are prognostic factors, a subsample consisting of participants reporting PFS at baseline will be selected. Subsequently, a predictive model will be made to assess which characteristics are associated to the course of (clusters of PFS) during follow-up. To explore whether sex- and gender-differences are present, we will perform most of the analyses separately for sex (male and female subjects). The main reason for this is that the questionnaires to measure PFS among women (female subjects) and men (male subjects) are different to each other. We would introduce bias if we would use the complete set of data and add sex as interaction term in the regression analyses. To explore the influence of gender-specific variables, we will add the gender identity variable and gender role variables in the regression analyses.

   Variables will be entered into the model using the ''enter'' method of regression (ie, all variables are forced into the model simultaneously, without making a decision about the order in which the variables are entered.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to participate in the observational prospective cohort study, when they are 16 years or older and don't meet any exclusion criteria.

Exclusion Criteria:

The general practices will perform the selection of potential participants.

A potential subject who meets any of the following criteria will not be invited for the prospective cohort study:

* terminal illnesses;
* cognitive impairment (e.g. due to dementia) precluding informed consent;
* current psychological condition precluding informed consent;
* not suitable or too ill to participate based on the judgement of the GP.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The cohort will be based on a community-dwelling population. The source population of the observational cohort study are people registered at a participating general practice.
Sampling Method: Probability Sample
Enrollment: 1691 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
sex- and gender differences in the prevalence of (clusters of) pelvic floor symptoms | prevalence at baseline
  To evaluate the sex-and gender difference in prevalence of (clinically relevant clusters of) PFS, the following primary parameters are assessed: lower urinary tract symptoms, bowel symptoms, prolapse, sexual functioning, and pain.
sex- and gender differences in the prevalence of (clusters of) pelvic floor symptoms | prevalence after 1 year
  To evaluate the sex-and gender difference in prevalence of (clinically relevant clusters of) PFS, the following primary parameters are assessed: lower urinary tract symptoms, bowel symptoms, prolapse, sexual functioning, and pain.
sex- and gender differences in the prevalence of (clusters of) pelvic floor symptoms | prevalence after 2 years
  To evaluate the sex-and gender difference in prevalence of (clinically relevant clusters of) PFS, the following primary parameters are assessed: lower urinary tract symptoms, bowel symptoms, prolapse, sexual functioning, and pain.
sex- and gender differences in the incidence of (clusters of) pelvic floor symptoms | after 1 year
  sex- and gender differences in the incidence of (clusters of) pelvic floor symptoms
sex- and gender differences in the incidence of (clusters of) pelvic floor symptoms | after 2 years
  sex- and gender differences in the incidence of (clusters of) pelvic floor symptoms

SECONDARY OUTCOMES:
risk factors | at baseline, after 1 year, after 2 years
  sex- and gender differences in the factors associated with the development of PFS
prognostic factors | at baseline, after 1 year, after 2 years
  sex- and gender differences in the factors that predict the course of PFS
impact of PFS on daily functioning | at baseline, after 1 year, after 2 years
  sex- and gender differences in the factors that reveal the impact of PFS on daily life
help seeking behavior | at baseline, after 1 year, after 2 years
  sex- and gender differences in help seeking behavior
health care use | at baseline, after 1 year, after 2 years
  sex- and gender differences in consultations for PFS and consultation frequency, diagnostic tests, diagnoses, treatment, and referrals

CONTACTS AND LOCATIONS:
Overall Officials: Marco H Blanker, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Notenboom-Nas FJM, Knol-de Vries GE, Beijer L, Tolsma Y, Slieker-Ten Hove MCP, Dekker JH, van Koeveringe GA, Blanker MH. Exploring pelvic floor muscle function in men with and without pelvic floor symptoms: A population-based study. Neurourol Urodyn. 2022 Nov;41(8):1739-1748. doi: 10.1002/nau.24996. Epub 2022 Jul 25. PMID 35876473